CLINICAL TRIAL: NCT03003312
Title: Prevalence of Pediatric Urolithiasis in Kashgar Area of Xinjiang in China: a Population and Ultrasonography Based Cross-sectional Study
Brief Title: Prevalence of Pediatric Urolithiasis in Kashgar Area of Xinjiang in China
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Guohua Zeng (Other)
Responsible Party: Sponsor-Investigator, Guohua Zeng, Vice-president, The First Affiliated Hospital of Guangzhou Medical University
Organization: The First Affiliated Hospital of Guangzhou Medical University (Other)
Other Study IDs: MRER(30)2016
Record Dates: First submitted 2016-10-27; First posted 2016-12-28 (Estimated); Last update posted 2016-12-28 (Estimated); Status verified 2016-11

CONDITIONS: Urolithiasis
Keywords: Urolithiasis; Uyghur; Prevalence; Associated factors; Children
MeSH Terms: conditions — Urolithiasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A blood sample of each child will be preserved in a -80℃refrigerator for further analysis of etiology of urolithiasis which include genetics.
Oversight: Data Monitoring Committee: No

SUMMARY:
Objective:The aim of this study is to investigate the prevalence and associated factors of pediatric urolithiasis in Kashgar area in China.

Methods: The investigators carry out a cross-sectional survey among children aged 0 to14 years across Kashgar area in China. The participants are selected by a two-stage and clustered random sampling method. Participants are asked to undergo urinary tract ultrasonographic examinations, provided blood and urine samples to analyze. Their parents or guardians are asked to fill out the questionnaires. Children those who are found with any abnormalities of their urinary system by ulrtasonography will undergo a low-dose computed tomography (CT) to confirm the abnormalities. The end point of this study is to calculate the prevalence rate, distribution and associated factors of pediatric urolithiasis in Kashi area.

DETAILED DESCRIPTION:
Background: Urolithiasis in children is a painful and costly disease that may also have detrimental long-term effects on kidney function. Although urolithiasis is rarely found in the pediatric population, several studies indicated that the incidence and inpatient hospitalization rates were sharply increased. The incidence of nephrolithiasis for children aged 18 years in South Carolina was 18.5 per 100,000 children in 2007, much higher than 7.9 per 100,000 in 1996. Data from Iceland revealed an incidence of 5.6 per 100,000 children aged 0 to 18 years on the basis of 26 new diagnoses of renal stone during a 6-year period among a national population of approximately 78,000 children. The composition analysis of stone in children revealed that the calcium stone was the most common one, accounted for 72% to 88%, and the uric acid stone accounted for 2% to 3% while the infective stone (included ammonium acid urate and magnesium ammonium phosphate) was rare.

Kashgar area lies in the southwest of Xinjiang province in China, with a climate of less annual rainfall, long hours of sunshine, high temperature and dry air. The population of Kashgar area is about 4 million and the Uighur residents account for about 90%.Pediatirc urolithiasis is a very common disease in Kashgar area. From August 2014 to July 2016, there were 708 pediatric patients with urolithiasis were treated in the department of urology in the First People's Hospital of Kashgar area which is a central hospital. The stone analysis of these pediatric patients by infrared spectroscopy indicated that ammonium acid urate accounted for 66%, magnesium ammonium phosphate accounted for 2.5%, uric acid accounted for 11%, and calcium stone accounted for 19% (these data has not been published ).This was very different from previous studies.

So we wonder urolithiasis maybe a very common disease among children in Kashgar area, even in south Xinjiang province. And maybe there are some special reasons for pediatric urolithiasis formation in this area.

Methods Study design and participants: A cross-sectional survey is carried out among children aged 0 to 14 years in Kashgar area in China. Before designed the study, we have conducted a pre-survey in a village which had 418 children by randomness clustered selected in Kashgar area. And ten children were found with urinary stone by ultrasonography. So we estimate the prevalence of pediatric urolithiasis (p) in this area is about 2.4% (10/418), with α of 0.05, a margin of error of less than 0.5%, 3599 children would needed by the formula of sample size caculation.Consider a relative sampling error of 10%, a predicted 20% refusal rate, and at least 4751 target children will be needed in this study.

Randomization: A two-stage and clustered random sampling method is used to select a representative sample of children across Kashgar area. The sampling process is initially stratified the 12 regions of Kashgar area (Kashi, Taxian, Shule, Zhepu, Yuepu, Bachu, Maigaiti, Yuecheng, Jiashi, Shufu, Shache, and Yingjisha) in descending order by Gross Domestic Product (GDP) 2014. The first tier is selected two regions by simple random sampling in the first six regions and the last six regions separately. Then the selected regions are stratified by the degree of urbanization (urban area vs rural area), and one community in urban area and one village in rural area is selected by randomization. At last four communities in urban area and four villages in rural area are selected across Kashgar area. Children those aged 0 to14 years in these selected communities and villages were all our target population.

Data collection:

The data include urinary tract ultrasonography (UTU), a standard questionnaire, urine examines and blood species. All of examinations are free of charge. All data are collected by investigators of our research group in community clinics of participant's residential area.

1. Appointment: After obtaining the population information from the local government, we will visit every family or household accompanied by staffs of the selected communities or villages, to obtain pediatric information of each family, explain the aim of the study, and invite the parents to take their kids to participate in the study which is held at the community of village clinic. Also we will give a notice that include the aim of the study, contents, date, and matter need attention of this survey to the parents.
2. Inform consent form: When the parents and children coming to the clinic, the investigators will explain the details of consent form to the parents again. If the parents are fully understand the aim of the study and agree to let their kids to participant in this study, they will be asked to sign their name and the date on the consent form. Also, the investigators will be required to sign the name and date on the same page.
3. Anthropometric indexes: Height (cm) and weight (kg) is measured using weighting-scale. Circumference of head, chest, arm and forearm is measured by a same tape. Subcutaneous fat thickness of triceps, biceps, scapular region, and abdominal wall is measured by a subcutaneous fat meter. All values are recorded on the first page of the questionnaire.
4. Blood specimen collecting and analysis: All children are invited to collect vein blood to analysis. The standard blood analysis protocol includes complete blood count (CBC), serum creatinine, urea, and uric acid. Blood samples for CBC analysis are collected using tubes with EDTA-K2 as preservative and are frozen at 4℃.Blood samples for serum chemistries analysis are collected using tubes without any preservative. All blood samples are delivered to the First People's Hospital of Kashgar area for analysis by automated analyzers. All blood samples are analyzed in 12 hours after collection. Also, we will preserve a blood sample of each child in a -80℃refrigerator for further analysis of etiology which include genetics.
5. Questionnaire: All parents are invited to fill out a pre-designed and standardized questionnaire by face to face interview of our Uygur staffs. Information on demographic data, feeding patterns, lifestyle, information of parents and family, possible symptoms of urinary stone, co-morbidities of kids, history of medicine, family history are recorded. Completeness and accuracy of questionnaires are checked up on site by special quality controller.
6. UTU: UTU is conducted by using same model of ultrasound machines with a 3.0-5.0 MHz frequency probe throughout this study. We will provide enough water to drink and all participants are required to have moderate bladder filling. Initially, participants lay in a prone position for scanning of bilateral kidneys and upper ureters. Then participants will turn to a supine position to have lower ureters and bladder scanned. The position is adjusted if necessary to achieve successful scanning. Details of the abnormalities are record including stone size, number, location, depth of hydronephrosis (mm). The longest axis of the stone in millimeter (mm) is used for the stone size. And also all the children which are found with urinary abnormalities are asked to undergo a Non-enhanced helical CT scans with two-mm slices in the First People's Hospital of Kashgar area.
7. Urine samples of children are collected after finishing UTU. All urine samples are analyzed by semi-automatic analyzers with dry chemical method on site.
8. Dietary record of case-control study: When one child is found with urinary stone, we will ask his/her parents to make a dietary record for three consecutive days by weight method. And also we will select four healthy children which have the same age and gender and ask their parents to make a dietary record with the same method. We will provide a weigh for each family. The table of dietary record is printed in Uygur.
9. Quality control: The investigators involved in this study have completed a training program on the methodology and data acquisition procedures. Each of them have a procedure manual that detailed the administration of the questionnaires, operation of the UTU, measurements of the anthropometric indexes, along with collecting and handling the blood specimens. The same doctor and machine of ultrasound is used during the whole study. All collected data will be registered and treated with the Epidata software (version 3.1).
10. End points evaluation: Prevalence is separately calculated for all participants and for their subgroups according to age, sex, urban or rural residence, BMI and family history of urinary stones, which is expressed as an unadjusted rate with 95% confidence intervals (CIs). Difference between the categorical variables is compared using the chi-square test. The association between urinary stone and relevant covariates is calculated using binary logistic regression models.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 0 to 14 years and live in Kashgar area in China.

Exclusion Criteria:

* Children aged 15 to 17 years live in Kashgar area in China.

Ages: 1 Day to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged 0 to 14 years live in Kashgar area in China.
Sampling Method: Probability Sample
Enrollment: 4751 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Prevalence of urolithasis among children in Kashgar area in Xinjiang, China. | From July 2016 to June 2017
  We are conducting a cross-sectional and ultrosound based survey among children aged 0 to 14 years across Kashgar area in China to evaluate the prevalence and associated factors of urolithiasis.This survey has been started in July 2016.

SECONDARY OUTCOMES:
The weight of children aged 0 to 14 years in Kashgar area in Xinjiang, China. | From July 2016 to June 2017
  We evaluate the development status of children in Kashgar according these anthropometric indexes: weight (kilogram) .
The development status of children aged 0 to 14 years in Kashgar area in Xinjiang, China. | From July 2016 to June 2017
  2、We evaluate the development status of children in Kashgar according these anthropometric indexes: height (centimeter)，circumference of head (centimeter), chest (centimeter), arm (centimeter), and forearm (centimeter).
The development status of children aged 0 to 14 years in Kashgar area. | From July 2016 to June 2017
  We evaluate the development status of children in Kashgar according these anthropometric indexes: subcutaneous fat thickness of triceps (millimeter), biceps (millimeter), scapular region (millimeter), and abdominal wall (millimeter).
Associated factors of urolithasis among children in Kashgar area in Xinjiang, China. | From July 2016 to June 2017
  We are conducting a cross-sectional and ultrosound based survey among children aged 0 to 14 years across Kashgar area in China to evaluate the prevalence and associated factors of urolithiasis.This survey has been started in July 2016.

OTHER OUTCOMES:
The nutrition status between children with urolithiassis and healthy kids. | From July 2016 to June 2017
  We also carry out a case-control study of comparing dietary nutrition between children with urolithiasis and healthy kids of 1:4. During the cross-sectional study, when one child is found with urinary stone, we will ask his/her parents to make a dietary record for three consecutive days by weight method. And also we will select four healthy children which have the same age and gender and ask their parents to make a dietary record with the same method.

CONTACTS AND LOCATIONS:
Overall Officials: Guohua Zeng, PH.D and M.D, Study Chair — The First Affiliated Hospital of Guangzhou Medical University
Locations (2):
- China (2):
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - The First People's Hospital of Kashgar Area, Kashgar, Xinjiang

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Penido MG, Tavares Mde S. Pediatric primary urolithiasis: Symptoms, medical management and prevention strategies. World J Nephrol. 2015 Sep 6;4(4):444-54. doi: 10.5527/wjn.v4.i4.444. PMID 26380196
- [Result] Clayton DB, Pope JC. The increasing pediatric stone disease problem. Ther Adv Urol. 2011 Feb;3(1):3-12. doi: 10.1177/1756287211400491. PMID 21789094
- [Result] Wang HH, Wiener JS, Lipkin ME, Scales CD Jr, Ross SS, Routh JC. Estimating the nationwide, hospital based economic impact of pediatric urolithiasis. J Urol. 2015 May;193(5 Suppl):1855-9. doi: 10.1016/j.juro.2014.09.116. Epub 2014 Oct 8. PMID 25305358
- [Result] Dwyer ME, Krambeck AE, Bergstralh EJ, Milliner DS, Lieske JC, Rule AD. Temporal trends in incidence of kidney stones among children: a 25-year population based study. J Urol. 2012 Jul;188(1):247-52. doi: 10.1016/j.juro.2012.03.021. Epub 2012 May 15. PMID 22595060